CLINICAL TRIAL: NCT01764893
Title: A Randomized, Double-Blind, Placebo-Controlled Study Assessing the Efficacy of Solifenacin and Percutaneous Tibial Nerve Stimulation in Patients With Refractory Overactive Bladder
Brief Title: Use of Percutaneous Tibial Nerve Stimulation With Solifenacin or Placebo to Treat Refractory Overactive Bladder
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Enrolling too slowly due to insurance plans no longer covering the cost of the Percutaneous Tibial Nerve Stimulation treatment.
Sponsor: Bay State Clinical Trials, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BSU-SOL-001
Record Dates: First submitted 2013-01-03; First posted 2013-01-10 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-05

CONDITIONS: Overactive Bladder
Keywords: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Solifenacin Succinate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PTNS and solifenacin (Active Comparator): PTNS bladder neuromodulation weekly for 12 treatments; solifenacin 5 mg capsule daily for 15 weeks
  Interventions: Other: PTNS plus solifenacin
- PTNS and placebo (Placebo Comparator): PTNS bladder neuromodulation weekly for 12 treatments; placebo 1 capsule daily for 15 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Other: PTNS plus solifenacin — 12 weekly treatments with percutaneous tibial nerve stimulation with 5 mg of solifenacin; an additional 4 weeks of solifenacin for a total of 15 weeks of study drug.
  Other Names: Vesicare
  Arms: PTNS and solifenacin
Other: Placebo — 12 weekly treatments with percutaneous tibial nerve stimulation with placebo; an additional 4 weeks of placebo for a total of 15 weeks of placebo.
  Arms: PTNS and placebo

SUMMARY:
The null hypothesis for this study is that the combination of solifenacin and Percutaneous Tibial Nerve Stimulation (PTNS) is not different from PTNS alone. However the investigators anticipate a 20% improvement in patients receiving combination therapy as measured by the OAB-q (Overactive Bladder questionnaire) scores.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. history of overactive bladder
3. history of inadequate response to prior or current treatment with anti- muscarinic medication, or unacceptable side effects from higher dose of anti-muscarinic medication
4. PTNS-naive
5. willing to discontinue the use of anti-muscarinic agents for 2 weeks before start of study medication ("washing out")
6. able to swallow and retain oral medication
7. able and willing to participate in the full duration of the study
8. able to read and write (health outcomes questionnaires are self-administered)and understand instructions related to study procedures and give written informed consent
9. OAB-q (items 1-8) score of 30 or higher

Exclusion Criteria:

1. presence of cardiac pacemaker and/or defibrillator
2. history of urinary retention
3. history of gastric retention
4. uncontrolled narrow angle glaucoma
5. any unstable, serious co-existing medical condition(s) including, but not limited to, myocardial infarction,coronary bypass surgery, unstable angina, cardiac arrhythmias, clinically evident congestive heart failure, or cerebrovascular accident within 3 months prior to Screening visit
6. abnormal liver function test (greater than 3 times the upper limit of normal for alanine aminotransferase [ALT], aspartate aminotransferase [AST], or alkaline phosphatase [ALP]); or bilirubin > 3 times the upper limit of normal
7. history of any illness (including psychiatric) that, in the opinion of the investigator, might confound the results of the study or pose additional risk to the subject
8. known hypersensitivity to solifenacin
9. participation in any investigational or marketed drug trial within the 30 days prior to the first dose of study drug or any time during the study period
10. pregnancy or trying to become pregnant
11. breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Overactive Bladder Questionnaire, items 1-8 only | Change from Baseline in Overactive Bladder Questionnaire at 11 weeks.
Overactive Bladder Questionnaire, items 1-8 only | Change from Baseline in Overactive Bladder Questionnaire at 15 weeks.

SECONDARY OUTCOMES:
3-day micturition diary | Change in Bladder diary from Baseline to 5 weeks.
  To measure changes in frequency, urgency, urge incontinence episodes, nocturia and urine volume (one day of each 3-day diary)
3-day micturition diary | Change in Bladder diary from Baseline to 11 weeks.
  To measure changes in frequency, urgency, urge incontinence episodes, nocturia and urine volume (one day of each 3-day diary)
3-day micturition diary | Change in Bladder diary from Baseline to 15 weeks.
  To measure changes in frequency, urgency, urge incontinence episodes, nocturia and urine volume (one day of each 3-day diary)
Urgency Perception Scale (questionnaire) | Changes in Urgency Perception from Baseline to 11 weeks.
Urgency Perception Scale (questionnaire) | Changes in Urgency Perception from Baseline to 15 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: H. David Mitcheson, MD, Principal Investigator — Bay State Clinical Trials, Inc.
Locations (1):
- Bay State Clinical Trials, Inc., Watertown, Massachusetts, United States